CLINICAL TRIAL: NCT05553353
Title: Evaluating a Novel Method to Determine the rTMS Dose Needed for Treating Depression After Spinal Cord Injury
Brief Title: Dosing rTMS for Depression Post-SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3972-W; 1IK2RX003972-01A1 (NIH)
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries; Depression; Depressive Disorder, Major
Keywords: Spinal Cord Injuries; Depression; Depressive Disorder, Major; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Depression; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Participants will:
  1. undergo high-resolution T1- and T2-weighted MRI scanning. These images will be used for image guided TMS assessments and e-field calculations for rTMS intensity.
  2. undergo rTMS to the left dorsolateral prefrontal cortex (DLPFC) as a treatment approach for depression. Treatment (active or sham) will be performed five times/week for six weeks (30 sessions). A total of 3,000 pulses/session will be delivered at 10Hz (4 seconds on and 26 seconds off) for a total of 75 stimulation cycles that lasts 37.5 minutes. The intensity will be individualized, as it will be based on reverse-calculation electric-field modeling. Participants receiving sham stimulation will undergo the same procedures as active rTMS except that a coil specifically designed to provide sham stimulation that is double-blinded will be utilized.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * Participants will be blinded to group (active vs. sham) assignments.
  * The assessor performing the resting motor threshold (rMT) testing will be blinded to any pre-determined electric-field modeling values or group assignments.
  * Staff member applying the rTMS treatment will be blinded, and an unblinded study staff member will set up the appropriate coil (active vs. sham) prior to each treatment session.
  * The staff member completing outcome assessments will be blinded to participant group assignments.
  * During the immediate post-testing session, the staff members applying the rTMS treatments and those completing the outcome assessments, as well as each participant, will be asked if they think active or sham treatment was received. This will allow for post-hoc assessment on blinding.
  * Unblinding will only occur in the case of a medical emergency or after all follow-up testing has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS (Experimental): Active repetitive transcranial magnetic stimulation (rTMS) that will be administered 5 days/week for 6 weeks. Intensity will be individualized based on reverse-calculation electric-field modeling.
  Interventions: Device: repetitive transcranial magnetic stimulation--Active
- Sham rTMS (Sham Comparator): Sham repetitive transcranial magnetic stimulation (rTMS) that will be administered 5 days/week for 6 weeks. Intensity will be individualized based on reverse-calculation electric-field modeling, but a sham treatment coil will be used; thus, no active treatment will be administered.
  Interventions: Device: repetitive transcranial magnetic stimulation--Sham

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation--Active — Repetitive transcranial magnetic stimulation (rTMS) is a type of non-invasive brain stimulation. An active coil will be used to administer the active rTMS.
  Other Names: rTMS
  Arms: Active rTMS
Device: repetitive transcranial magnetic stimulation--Sham — Repetitive transcranial magnetic stimulation (rTMS) is a type of non-invasive brain stimulation. A sham coil will be used to administer the sham rTMS.
  Other Names: rTMS
  Arms: Sham rTMS

SUMMARY:
Depression is a leading cause of disability worldwide and is more commonly seen in individual's post-spinal cord injury (SCI) than in the general population. Depression post-SCI impacts an individuals' quality of life and recovery. It has been reported that among Veterans with an SCI, those without depression live longer than those with depression. Thus, depression must be treated appropriately. Repetitive transcranial magnetic stimulation (rTMS) is an FDA-approved treatment for depression, but dosing is based on a motor response or movement in the thumb. Over half of individuals with SCI have some degree of arm or hand impairment, so these individuals might not be eligible for rTMS, or they may receive the wrong dose. This study proposes clinical trial in individuals with depression post-SCI to assess the anti-depressant effect of a novel technique to dose rTMS that does not require a motor response in the thumb. By gaining a better understanding of the application of rTMS for depression post-SCI, the investigators aim to advance the rehabilitative care of Veterans.

DETAILED DESCRIPTION:
Depression is a leading cause of disability worldwide and is one of the most prevalent neuropsychiatric manifestations following spinal cord injury (SCI). Based on an estimated 42,000 Veterans having an SCI1 and an estimated prevalence of depression among Veterans post-SCI of 19-28%, nearly 12,000 Veterans with SCI have comorbid depression at any time. The burden of depression post-SCI is significant, as it can impact quality of life and is associated with increased healthcare utilization and higher mortality. As noted by the updated Clinical Practice Guidelines from the Paralyzed Veterans of America, treating depression is essential, but further research is needed specifically within the SCI population to help formulate stronger evidence-based guidelines.

Repetitive transcranial magnetic stimulation (rTMS), a type of non-invasive brain stimulation, is an FDA-approved treatment option for major depressive disorder (MDD) that is utilized throughout the Veterans Affairs (VA) health system. However, to date, no published studies have examined its effectiveness post-SCI. A critical challenge for widespread administration of rTMS for depression post-SCI is dosing, as the resting motor threshold (rMT), a motor response to transcranial magnetic stimulation (TMS), of the right abductor pollicis brevis (APB) is used to dose rTMS. Approximately 60% of the SCI population has incomplete or complete tetraplegia, indicating some degree of upper extremity (UE) impairment, making rMT not reliably attainable. Thus, it is plausible to conclude that over half the SCI population could be excluded from receiving rTMS treatment for depression or may receive an improper dose, impacting its safety and effectiveness. This represents a major gap in the field of SCI rehabilitation in that a large portion of individuals with SCI have concurrent MDD. As such, evidence-based treatment options are necessary to address the needs of this large clinical cohort, thereby improving the lives of these Veterans, their caregivers, and their families.

This study will examine the potential of rTMS, dosed by reverse-calculation electric-field modeling, to improve depressive symptoms in individuals with MDD post-SCI via a randomized, 2-arm, sham-controlled pilot clinical trial. Over four years, twenty-four individual post-SCI with MDD will be enrolled and randomized to receive 6 weeks (5 sessions/week) of either active or sham rTMS treatment. Using an unbalanced design, a quarter of the sample (n=6) randomized to the sham group and the remainder (n=18) randomized to receive active rTMS. Dosing parameters will follow the FDA-approved protocol of 3,000 pulses/session at 10Hz, and intensity will be determined by reverse-calculation electric-field modeling. The primary outcome measure for this study will be the Hamilton Rating Scale for Depression-17. Participants will also complete a 12- and 24-week post-intervention follow-up assessments. It is hypothesized that rTMS treatment dosed using reverse-calculation electric-field modeling will result in a moderate between-group effect size favoring the anti-depressant benefits of rTMS treatment (vs. sham).

In addition to its established anti-depressive effects, rTMS has also been shown to improve patient-reported outcomes such as quality of life and depression-related disability. An extremely exciting possibility is that effective treatment of MDD results in a virtuous cycle whereby reducing depression concomitantly facilitates improvements in other psychosocial domains. The second aim seeks to explore this possibility by determining the extent to which improvements in depressive symptoms are associated with changes in quality of life and participation in Veterans post-SCI with MDD. This trial is an essential step toward optimizing SCI rehabilitation, while simultaneously providing a unique opportunity to study the effects of depression on psychosocial responses to rehabilitation.

The data generated could inform the development of additional interventions focused on neuromodulation to improve function and quality of life for individuals following SCI and other clinical cohorts with upper extremity motor impairment, (e.g., traumatic brain injury, multiple sclerosis, amputees) who otherwise may not be able to benefit from the anti-depressant effects of rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

* cervical or thoracic spinal cord injury at least 6 months prior with AIS A, B, C, or D;
* 18 - 60 years of age;
* major depressive disorder, as identified by Structured Clinical Interview for DSM-V;
* Hamilton Depression Rating Scale-17 score > 18;
* not taking antidepressant medications or no change in doses of psychotropic medication(s) for at least 4 weeks before the study (6 weeks if newly initiated medication)

Exclusion Criteria:

* concomitant neurologic diseases/disorders or dementia;
* cognitive impairment (Montreal Cognitive Assessment <17);
* history of psychosis or other Axis I disorder that is primary;
* positive screen for bipolar disorder through the Mini-International Neuropsychiatric Interview;
* history of claustrophobia;
* life expectancy <1 year;
* electronic or metallic implants (i.e., metal in the head, cochlear implant, or pacemaker;
* history of seizures or currently prescribed anti-seizure medications;
* taking medication that increases the risk of seizures;
* pregnancy as identified through a positive urine pregnancy test;
* Hamilton Depression Rating Scale-17 question #3 regarding suicide: >2 or suicide attempt within the previous two years;
* inability to (University of California, San Diego Brief Assessment of Capacity to Consent) or declined to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Rating Scale-17 (HAM-D17) score immediately post-intervention | Baseline; Following Week 2 of 6-week intervention Following Week 4 of 6-week intervention; Immediately post-intervention; 12-weeks post-intervention; 24-weeks post-intervention
  The Hamilton Rating Scale for Depression (HAM-D17) is the most widely used tool to assess the severity of depressive symptoms, once diagnosed, and will be used in this study. The HAM-D17 is a semi-structured interview style questionnaire that asks about one's experience with seventeen different depressive symptoms over the past week. Total HAM-D17 scores range from no depressive symptoms (HAM-D17 = 0-7); mild (HAM-D17 = 8-16), moderate (HAM-D17 = 17-23) or severe depressive symptoms (HAMD-D17 = 24).

SECONDARY OUTCOMES:
Change from baseline in Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) at timepoints noted below | Baseline; Following Week 2 of 6-week intervention Following Week 4 of 6-week intervention; Immediately post-intervention; 12-weeks post-intervention; 24-weeks post-intervention
  The Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF) is a 16-item questionnaire that asks about the degree of enjoyment and satisfaction in various are of daily functioning, like physical health/activity, mood, work, household duties, school/coursework, leisure time activity, and social relationships. Answers are scored from 1 (very poor) to 5 (very good). It is a valid and reliable measure often used in psychiatric research but has been used in SCI research for neuropathic pain.
Change from baseline in Sheehan Disability Scale (SDS) Score at timepoints noted below | Baseline; Following Week 2 of 6-week intervention Following Week 4 of 6-week intervention; Immediately post-intervention; 12-weeks post-intervention; 24-weeks post-intervention
  Sheehan Disability Scale (SDS): The SDS is a three-item questionnaire that asks how depressive symptoms have impacted work/school, social, and family. It is based on a 10-point scale, where 0 = no disruption to 10 = extreme disruption. This outcome use used in the only randomized control trial for an antidepressant post-SCI.
Change from baseline in Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) Score at timepoints noted below | Baseline; Following Week 2 of 6-week intervention Following Week 4 of 6-week intervention; Immediately post-intervention; 12-weeks post-intervention; 24-weeks post-intervention
  Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI) is used to assess physical activity levels of individuals with a spinal cord injury. This is a 3-item questionnaire that asks one to report the number of days and minutes of mild, moderate, and heavy-intensity leisure-time physical activity performed over the previous seven days. This is a valid and reliable measure in the SCI population.
Change from baseline in Craig Handicap Assessment and Reporting Tool - Short Form (CHART-SF) Score at timepoints noted below | Baseline; Following Week 2 of 6-week intervention Following Week 4 of 6-week intervention; Immediately post-intervention; 12-weeks post-intervention; 24-weeks post-intervention
  Craig Handicap Assessment and Reporting Tool - Short Form (CHART-SF) assesses how an individual with a disability fulfills roles in six domains, physical independence, cognitive independence, mobility, occupation, social integration, and economic self-sufficiency. It is a valid and reliable measure post-spinal cord injury. The total score ranges from 0 - 600, with a higher score indicating greater independent functioning and higher social and community participation.
Change from baseline in Reintegration to Normal Living Index (RNL) Score at timepoints noted below | Baseline; Following Week 2 of 6-week intervention Following Week 4 of 6-week intervention; Immediately post-intervention; 12-weeks post-intervention; 24-weeks post-intervention
  The Reintegration to Normal Living Index (RNL) is an 11-item questionnaire that assesses one's satisfaction with their performance of mobility, self-care, daily activity, recreational activity, and family roles. The total adjusted score ranging from 0 - 100, with 100 indicating full or complete reintegration.
Change from baseline Hamilton Depression Rating Scale-17 (HAM-D17) Score at timepoints noted below | Baseline; Following Week 2 of 6-week intervention Following Week 4 of 6-week intervention; 12-weeks post-intervention; 24-weeks post-intervention
  The Hamilton Rating Scale for Depression (HAM-D17) is the most widely used tool to assess the severity of depressive symptoms, once diagnosed, and will be used in this study. The HAM-D17 is a semi-structured interview style questionnaire that asks about one's experience with seventeen different depressive symptoms over the past week. Total HAM-D17 scores range from no depressive symptoms (HAM-D17 = 0-7); mild (HAM-D17 = 8-16), moderate (HAM-D17 = 17-23) or severe depressive symptoms (HAMD-D17 = 24).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J VanDerwerker, PhD DPT PT, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No